CLINICAL TRIAL: NCT00527098
Title: Optimal Fluid Resuscitation for Trauma Patients
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kenneth Proctor, Professor, University of Miami
Other Study IDs: 20070108
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Results first posted 2011-05-04 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Trauma
Keywords: Trauma Resuscitation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if the overall fluid requirements for the first 24 hours after admission will be reduced with Hextend versus a standard of care crystalloid resuscitation fluid.

DETAILED DESCRIPTION:
Following severe multi-system traumatic injury, the first 24 hours of standard resuscitation fluid will be either Hextend or crystalloid depending upon attending preference. No tests or interventions will be performed for research purposes.

Data will be collected prospectively from patient medical records and attending clinicians to monitor fluid requirements, hemodynamics and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years old and less than 65 years old
* Admission with multi-system traumatic injury
* Admission to the intensive care unit

Exclusion Criteria:

* Less than 18 or greater than 65 years old
* Pregnant or lactating
* No fluid resuscitation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Trauma Patients
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Proctor, PhD, Principal Investigator — University of Miami; Carl I Schulman, MD, MSPH, Study Director — University of Miami
Locations (1):
- Ryder Trauma Center, Miami, Florida, United States

REFERENCES:
- [Background] Earle SA, de Moya MA, Zuccarelli JE, Norenberg MD, Proctor KG. Cerebrovascular resuscitation after polytrauma and fluid restriction. J Am Coll Surg. 2007 Feb;204(2):261-75. doi: 10.1016/j.jamcollsurg.2006.11.014. PMID 17254930
- [Background] Crookes BA, Cohn SM, Bonet H, Burton EA, Nelson J, Majetschak M, Varon AJ, Linden JM, Proctor KG. Building a better fluid for emergency resuscitation of traumatic brain injury. J Trauma. 2004 Sep;57(3):547-54. doi: 10.1097/01.ta.0000135162.85859.4c. PMID 15454801
- [Background] King DR, Cohn SM, Proctor KG. Changes in intracranial pressure, coagulation, and neurologic outcome after resuscitation from experimental traumatic brain injury with hetastarch. Surgery. 2004 Aug;136(2):355-63. doi: 10.1016/j.surg.2004.05.011. PMID 15300202
- [Background] Kelly ME, Miller PR, Greenhaw JJ, Fabian TC, Proctor KG. Novel resuscitation strategy for pulmonary contusion after severe chest trauma. J Trauma. 2003 Jul;55(1):94-105. doi: 10.1097/01.TA.0000029042.37577.A6. PMID 12855887

RESULTS

PARTICIPANT FLOW:
Groups:
- Hextend Plus Standard of Care: Hextend along with the routine Standard of Care Resuscitation Fluid
- Standard of Care: Routine Standard of Care Resuscitation Fluid
Period: Overall Study
Arm/Group | Hextend Plus Standard of Care | Standard of Care
Started | 36 | 83
Completed | 36 | 83
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hextend Plus Standard of Care | Standard of Care | Total
Number analyzed (Participants) | 36 | 83 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 83 | 119
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39 (17) | 39 (17) | 39 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 17 | 24
  Male | 29 | 66 | 95
Region of Enrollment [Number; unit: participants]
  United States | 36 | 83 | 119

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Time Frame: From hospital arrival up to an average of 3.5 weeks
Population: Analysis was per protocol.
Measure: Number; unit: participants
Groups:
- Observational: This is an observational trial.
Arm/Group | Observational
Number analyzed (Participants) | 119
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this observational study.
Arm/Group | Hextend Plus Standard of Care | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/83
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No